CLINICAL TRIAL: NCT05288673
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of ALXN1210 Administered Intravenously to Healthy Subjects
Brief Title: A Study of Multiple Doses of ALXN1210 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: ALXN1210-HV-102; 2014-005495-29 (EudraCT Number)
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: ALXN1210; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and on-site medical/nursing staff at the study site were blinded to study drug/dose assignment. The pharmacy staff who prepared ALXN1210 or placebo, however, was not blinded to study drug assignment, but all other site staff, including the Investigator and personnel administering study drug, was blinded. Sponsor staff was unblinded as needed (for example, to monitor the pharmacy), but did not share any information on study drug assignment with the site staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ALXN1210 400 mg (Experimental): Participants received ALXN1210 every 28 days.
  Interventions: Drug: ALXN1210
- ALXN1210: 800 mg (Experimental): Participants received ALXN1210 every 28 days.
  Interventions: Drug: ALXN1210
- Placebo (Placebo Comparator): Participants received placebo every 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN1210 — ALXN1210 was administered by IV infusion over 5 periods, 1 dose per period: Period 1, induction; Periods 2-5, maintenance. Participants received a total of 5 doses of 400 or 800 mg, each administered every 28 days.
  Other Names: Ultomiris; Ravulizumab
  Arms: ALXN1210 400 mg; ALXN1210: 800 mg
Drug: Placebo — Placebo was administered by IV infusion over 5 periods, 1 dose per period. Participants received the same volume and infusion rate as specified for each ALXN1210 dose (400 or 800 mg).
  Arms: Placebo

SUMMARY:
This study evaluated the safety and tolerability of multiple doses of ALXN1210 (400 and 800 milligrams [mg]) following intravenous (IV) administration to healthy participants.

DETAILED DESCRIPTION:
Participants were divided into 2 cohorts and were randomly assigned in a 3:1 ratio to receive IV ALXN1210 or placebo. Participants in Cohort 1 received 5 IV doses of 400 mg of ALXN1210 or placebo administered every 28 days. To determine if dose continuation and dose escalation to Cohort 2 should occur, the Safety Review Committee conducted a blinded review of the available safety data after Day 15 of the second dose of the last participant in Cohort 1. Participants in Cohort 2 received 5 doses of 400 mg of ALXN1210 or placebo and 5 IV doses of 800 mg of ALXN1210 or placebo administered intravenously every 28 days. Safety, PK, PD, and immunogenicity assessments were performed during the Follow-up Period after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants ≥ 25 and ≤ 55 years old; smokers (no more than 10 cigarettes daily), former smokers (at the Investigator's discretion), or nonsmokers.
* Body mass index from 18 through 29.9 kilogram (kg)/square meter, inclusive, and weight between 50 and 100 kg, inclusive.
* QT interval (corrected using the Fridericia formula) ≤ 450 milliseconds (ms) for males and ≤ 470 ms for females at Screening and prior to dosing on Day 1.
* Participant was willing and able to give written informed consent and comply with the study visit schedule.
* Documented vaccination with tetravalent meningococcal conjugate vaccine (MCV4) at least 56 days and not more than 3 years prior to dosing. Documentation must have included a positive serum bactericidal antibody test to confirm an immune response before the study drug administration.
* Vaccination with serogroup B vaccine at least 56 days prior to dosing on Day 1, with a booster administered at least 28 days prior to dosing on Day 1.
* Male participants with a female spouse/partner of childbearing potential or a pregnant or breastfeeding spouse or partner were required to use barrier contraception (male condom) during the treatment period and for at least 6 months after the last dose of ALXN1210.

Exclusion Criteria:

* Participants who had intimate and prolonged contact (defined as living under the same roof or providing personal care) with individuals who were either immunocompromised, or had specific underlying medical conditions (persons with anatomic or functional asplenia [including sickle cell disease]; persons with congenital complement, properdin, factor D, or primary antibody deficiencies, persons with acquired complement deficiencies [for example, those receiving eculizumab], and persons with human immunodeficiency virus [HIV]) or with persons younger than 2 years of age or older than 65 years of age
* Participants who were one of the following: professionals exposed to environments of greater risk for meningococcal disease; research, industrial, and clinical laboratory personnel routinely exposed to Neisseria meningitidis; military personnel during recruit training (military personnel may be at increased risk when accommodated in close quarters); daycare center workers; those living on a college or university campus; or those who planned to travel during the course of the study to or had travelled to endemic areas for meningococcal meningitis (for example, India, Sub-Saharan Africa, pilgrimage to Saudi Arabia for Hajj) within the past 6 months
* History of any Neisseria infection
* History of unexplained recurrent infection or infection that required treatment with systemic antibiotics within the last 90 days prior to dosing
* HIV infection (evidenced by HIV-1 or HIV-2 antibody titer)
* Acute or chronic hepatitis B virus infection (evidenced by the presence of hepatitis B surface antigen or immunoglobulin M antibodies against hepatitis B core antigen)
* Acute or chronic hepatitis C virus infection (evidenced by antibody titer)
* Active systemic viral or fungal infection within 14 days prior to dosing
* Positive or indeterminate QuantiFERON-TB test indicating possible tuberculosis infection
* History of latent or active tuberculosis or exposure to endemic areas within 8 weeks prior to the screening visit
* Female participants who were breastfeeding or were of childbearing potential, including any female who had experienced menarche and who had not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who was pregnant, breastfeeding, or not postmenopausal.
* Positive serum pregnancy test at Screening or Day -1
* Serum creatinine > upper limit of normal (ULN) of the reference range of the testing laboratory at Screening or Day -1.
* Alanine aminotransferase or aspartate aminotransferase > ULN of the reference range of the testing laboratory at Screening or > 1.5*ULN of the reference range of the testing laboratory at Day -1.
* Any of the following hematology results: hemoglobin < 135 grams (g)/L for males and < 120 g/L for females; hematocrit < 0.41 L/L for males and < 0.36 L/L for females; white blood cells < 3.5*10^3/microliter (μL) or > ULN of the testing laboratory reference range; absolute neutrophils < 1.5*10^3/μL (< 1.0*10^3/μL for black race participants) or > ULN of the testing laboratory reference range; and platelets < the lower limit of normal of the testing laboratory reference range or > 450*10^3/μL at Screening or Day -1; or complete blood count clinical laboratory results considered as clinically relevant and unacceptable by the Investigator at Day -1.
* History of complement deficiency or complement activity below normal reference range as evaluated by complement alternative pathway enzyme-linked immunosorbent assay at Screening.
* History of malignancy, other than basal cell carcinoma that had been treated and had no evidence of recurrence.
* Participation in a clinical study within 30 days before initiation of dosing on Day 1 or use of any experimental small-molecule therapy within 30 days prior to dosing on Day 1.
* Participation in more than 1 clinical study of a monoclonal antibody (mAb) or participation in a clinical study of a mAb within the 12 months prior to Screening during which the participant was exposed to the active study drug. Participants who had participated in only 1 study of an mAb were considered for enrollment if they had completed that study more than 12 months prior to Screening.
* Major surgery or hospitalization within 90 days prior to dosing.
* Contraindication to receiving MCV4 and/or serogroup B vaccine, including severe (life-threatening) allergic reaction to a previous dose of MCV4 and/or serogroup B vaccine, severe (life-threatening) allergy to any vaccine component, or previous diagnosis of Guillain-Barré syndrome.
* History of allergy to excipients of ALXN1210 (that is, polysorbate 80).
* Documented history of allergy to penicillin or cephalosporin.
* History of significant allergic reaction (anaphylaxis, angioedema) to any product (food, pharmaceutical, etc).
* Positive urine drug toxicology screen at Screening or Day -1.
* Donation of plasma within 7 days prior to dosing. Donation or loss (excluding volume drawn at Screening) of more than 50 mL of blood within 30 days of dosing or more than 499 mL of blood within 56 days of dosing.
* Use of prescription medications within 28 days prior to study drug administration.
* Clinical diagnosis of any autoimmune or rheumatologic disease (for example, systemic lupus erythematosus, rheumatoid arthritis).
* Immunization with a live-attenuated vaccine 1 month prior to dosing or planned vaccination during the course of the study (except for the vaccination planned by the study protocol).
* Presence of fever (confirmed body temperature > 37.6°C; for example, a fever associated with a symptomatic viral or bacterial infection) within 14 days prior to the first dose.
* Participants with any medical history, conditions or risks that, in the opinion of the Investigator, would have interfered with the participant's full participation in the study or compliance with the protocol, posed any additional risk for the participant, or confounded the assessment of the participant or outcome of the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: ALXN1210 400 mg: Participants received multiple doses of ALXN1210 400 milligrams (mg), via intravenous (IV) infusion on Day 1 and then every 28 days (Days 29, 57, 85, and 113) for a total of 4 doses. Participants were followed for 196 days.
- Cohort 2: ALXN1210 800 mg: Participants received multiple doses of ALXN1210 800 mg, via IV infusion on Day 1 and then every 28 days (Days 29, 57, 85, and 113) for a total of 4 doses. Participants were followed for 196 days.
- Placebo: Pooled: Participants received multiple doses of placebo matched to ALXN1210 400 mg or 800 mg, via IV infusion on Day 1 and then every 28 days (Days 29, 57, 85, and 113) for a total of 4 doses. Participants were followed for 196 days.
Period: Overall Study
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled
Started | 6 | 6 | 4
Received At Least 1 Dose Of Study Drug | 6 | 6 | 4
Completed | 6 | 6 | 3
Not Completed | 0 | 0 | 1
Not completed — Consent withdrawn by subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of ALXN1210 or placebo.
Groups:
- Cohort 1: ALXN1210 400 mg: Participants received multiple doses of ALXN1210 400 mg, via IV infusion on Day 1 and then every 28 days (Days 29, 57, 85, and 113) for a total of 4 doses. Participants were followed for 196 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled | Total
Number analyzed (Participants) | 6 | 6 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (4.32) | 35.2 (5.78) | 33.5 (8.70) | 32.3 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 6 | 4 | 16
Race/Ethnicity, Customized [Number; unit: Participants] — Number of participants based on race.
  Participants
    Not Hispanic or Latino | 6 | 6 | 4 | 16
Race/Ethnicity, Customized [Number; unit: Participants] — Number of participants based on ethnicity.
  Participants
    Black or African American | 2 | 0 | 1 | 3
    White | 4 | 6 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (for example, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or procedure, whether or not considered related to the medicinal product or procedure, which occurred during the course of the clinical study. TEAEs were defined as AEs that occurred on or after the date and time of study drug administration, or those that first occurred before dosing but worsened in frequency or severity after study drug administration. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Day 309
Population: The safety population consisted of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled
Number analyzed (Participants) | 6 | 6 | 4
Participants | 6 | 6 | 4

2. Secondary Outcome: Area Under The Serum Concentration Versus Time Curve From Time Zero To Infinity (AUCinf) of ALXN1210
Description: Blood samples were collected for estimation of AUCinf by noncompartmental analyses using Phoenix WinNonlin 6.3 or higher.
Time Frame: Predose, end of infusion, 30 minutes, 4 hours, 8 hours and 24 hours post start of infusion on Day 1 up to Day 309
Population: The pharmacokinetic (PK) population consisted of all participants who had sufficient serum concentration data to enable the calculation of PK parameters. Here, Number of Participants analyzed signifies those participants who were evaluable for this outcome measure. Data was collected from the cohorts treated with ALXN1210 only for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: hours*micrograms/milliliter (h*ug/mL)
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg
Number analyzed (Participants) | 6 | 5
hours*micrograms/milliliter (h*ug/mL) | 209047.941 (34101.040) | 489692.330 (58968.554)

3. Secondary Outcome: Area Under The Serum Concentration From Time Zero To The Time of The Last Quantifiable Concentration (AUCt) of ALXN1210
Description: Blood samples were collected for estimation of AUCt by noncompartmental analyses using Phoenix WinNonlin 6.3 or higher.
Time Frame: Predose, end of infusion, 30 minutes, 4 hours, 8 hours and 24 hours post start of infusion on Day 1 up to Day 309
Population: The PK population consisted of all participants who had sufficient serum concentration data to enable the calculation of PK parameters. Here, Number of Participants analyzed signifies those participants who were evaluable for this outcome measure. Data was collected from the cohorts treated with ALXN1210 only for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg
Number analyzed (Participants) | 6 | 5
h*ug/mL | 205241.063 (32514.529) | 478063.379 (54295.251)

4. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of ALXN1210
Description: Blood samples were collected for estimation of Cmax by noncompartmental analyses using Phoenix WinNonlin 6.3 or higher.
Time Frame: Predose, end of infusion, 30 minutes, 4 hours, 8 hours and 24 hours post start of infusion on Day 1 up to Day 309
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg
Number analyzed (Participants) | 6 | 5
ug/mL | 210.333 (34.869) | 454.400 (50.639)

5. Secondary Outcome: Percent Change From Baseline in Free Complement Protein C5 Concentration at Day 113
Description: Blood samples were collected for analysis of free C5 concentration.
Time Frame: Baseline, Day 113
Population: The pharmacodynamic (PD) population consisted of all participants who had sufficient total and/or free C5 concentration data, chicken red blood cells (cRBC) hemolysis data, or other data measuring C5 activation to enable the evaluation of the PD effects. Here, Number of Participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled
Number analyzed (Participants) | 6 | 5 | 4
Percent Change | -31.63 (15.484) | -93.8820 (11.2938) | -22.16 (15.965)

6. Secondary Outcome: Percent Change From Baseline in Total C5 Concentration at Day 113
Description: Blood samples were collected for analysis of total C5 concentration.
Time Frame: Baseline, Day 113
Population: The PD population consisted of all participants who had sufficient total and/or free C5 concentration data, cRBC hemolysis data, or other data measuring C5 activation to enable the evaluation of the PD effects. Here, Number of Participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled
Number analyzed (Participants) | 6 | 5 | 4
Percent Change | 42.57 (28.445) | 154.36 (23.053) | -8.65 (17.351)

7. Secondary Outcome: Percent Change From Baseline in Chicken Red Blood Cell Hemolysis at Day 113
Description: Blood samples were collected for analysis of cRBC hemolysis.
Time Frame: Baseline, Day 113
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled
Number analyzed (Participants) | 6 | 5 | 4
Percent Change | -52.53 (22.740) | -77.75 (28.579) | -7.28 (21.259)

8. Secondary Outcome: Percent Change From Baseline in C5 Activation at Day 113
Description: Blood samples were collected for analysis of C5 activation. Results are reported as percent change in both the complement classical pathway (CCP) activity response and the complement alternative pathway (CAP) activity response.
Time Frame: Baseline, Day 113
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled
Number analyzed (Participants) | 6 | 5 | 4
Percent Change
  CCP | -1.66 (6.049) | -15.16 (22.731) | 5.51 (10.839)
  CAP | -17.54 (18.849) | -39.76 (10.214) | -5.90 (16.896)

9. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADAs) to ALXN1210
Description: Blood samples were collected to evaluate antibody response through development of ADAs.
Time Frame: Baseline up to Day 309
Population: The immunogenicity analysis population consisted of all participants who had a pre-dose and post-dose ADA sample collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled
Number analyzed (Participants) | 6 | 6 | 4
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Day 309
Description: The safety population consisted of all participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1: ALXN1210 400 mg | Cohort 2: ALXN1210 800 mg | Placebo: Pooled
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ALXN1210 400 mg (N=6) | Cohort 2: ALXN1210 800 mg (N=6) | Placebo: Pooled (N=4)
Seasonal allergy (Immune system disorders) | 1 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 2 (7) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 3 (5) | 2 (4)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 2 (3)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes